CLINICAL TRIAL: NCT00103662
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Comparative Trial of AMD3100 Plus G-CSF Versus G-CSF Plus Placebo to Mobilize and Collect ≥ 6*10^6 CD34+ Cells/kg in Multiple Myeloma Patients for Autologous Transplantation
Brief Title: Mobilization of Stem Cells With AMD3100 (Plerixafor) in Multiple Myeloma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMD3100-3102; 2005-003599-39 (EudraCT Number); NCT00248417 (obsolete NCT alias)
Record Dates: First submitted 2005-02-11; First posted 2005-02-14 (Estimated); Results first posted 2010-09-29 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Granulocyte Colony-Stimulating Factor; plerixafor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- G-CSF plus plerixafor (Experimental)
  Interventions: Drug: Granulocyte colony-stimulating factor plus plerixafor
- G-CSF plus placebo (Placebo Comparator)
  Interventions: Drug: Granulocyte colony-stimulating factor plus placebo

INTERVENTIONS:
Drug: Granulocyte colony-stimulating factor plus plerixafor — Participants underwent mobilization with granulocyte colony-stimulating factor (G-CSF) (10 µg/kg/day) for 4 days, administered by subcutaneous (SC) injection. On the evening of Day 4, participants received plerixafor (240 µg/kg), administered by SC injection. On Day 5, participants received a morning dose of G-CSF (10 µg/kg) and underwent apheresis approx. 10 to 11 hours after the dose of plerixafor (within 60 minutes of G-CSF administration). Participants continued to receive an evening dose of plerixafor followed by a morning dose of G-CSF and apheresis for up to 4 aphereses or until ≥ 6*10^6 CD34+ cells/kg were collected. Participants who participated in the rescue procedure underwent an additional daily treatment with plerixafor (240 µg/kg) and apheresis for up to 4 days.
  Other Names: Mozobil; AMD3100
  Arms: G-CSF plus plerixafor
Drug: Granulocyte colony-stimulating factor plus placebo — Participants underwent mobilization with granulocyte colony-stimulating factor (G-CSF) (10 µg/kg/day) for 4 days, administered by subcutaneous (SC) injection. On the evening of Day 4, participants received placebo, administered by SC injection. On Day 5, participants received a morning dose of G-CSF (10 µg/kg) and underwent apheresis approx. 10 to 11 hours after the dose of placebo (within 60 minutes of G-CSF administration). Participants continued to receive an evening dose of placebo followed by a morning dose of G-CSF and apheresis for up to 4 aphereses or until ≥ 6*10^6 CD34+ cells/kg were collected. Participants who participated in the rescue procedure underwent an additional daily treatment with plerixafor (240 µg/kg) and apheresis for up to 4 days.
  Arms: G-CSF plus placebo

SUMMARY:
The purpose of this study is to determine whether the combination of AMD3100 (plerixafor) and granulocyte colony-stimulating factor (G-CSF, generic name of filgrastim) is better than G-CSF alone to mobilize and collect the optimal number of stem cells in multiple myeloma patients for autologous transplantation.

DETAILED DESCRIPTION:
A peripheral stem cell transplant may be able to replace blood-forming cells that were destroyed by chemotherapy. Currently filgrastim (G-CSF), a colony stimulating factor, is used to cause the growth and mobilization of stem cells from bone marrow to peripheral blood, which can then be collected from the peripheral blood by a process called apheresis. Plerixafor aids in the release of the stem cells from the bone marrow into the peripheral blood, possibly allowing for a more rapid collection of a larger number of stem cells from the peripheral blood. Larger stem cell doses for transplantation correlate to faster recovery times after high dose chemotherapy followed with stem cell transplantation. This study is intended to determine whether the combination of plerixafor with filgrastim (G-CSF)is better than filgrastim (G-CSF) alone in helping multiple myeloma patients collect at least 6 million stem cells in two or less apheresis sessions.

This study was previously posted by AnorMED, Inc. In November 2006, AnorMED, Inc. was acquired by Genzyme Corporation. Genzyme Corporation is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma in first or second complete or partial remission
* >= 4 weeks since last cycle of chemotherapy (thalidomide, dexamethasone, and Velcade were not considered prior chemotherapy for the purpose of this study)
* Recovered from all acute toxic effects of prior chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* White Blood Cell count (WBC) > 2.5*10^9/L
* Absolute polymorphonuclear leukocytes (PMN) count > 1.5*10^9/L
* Platelet (PLT) > 100*10^9/L
* Serum creatinine <=2.2 mg/dL
* Cardiac and pulmonary status sufficient to undergo apheresis and transplantation
* Negative for HIV

Exclusion Criteria):

* Failed previous stem cell collection
* Previous stem cell transplantation
* Brain metastases or myelomatous meningitis
* Radiation to ≥ 50% of the pelvis
* Abnormal electrocardiogram (ECG) with rhythm disturbance (ventricular arrhythmias) or other conduction abnormality
* Received bone-seeking radionuclides (e.g. holmium)
* A residual acute medical condition resulting from prior chemotherapy

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2005-01; Primary Completion 2006-10 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (39):
- United States (37):
  - City of Hope Samaritan Bone Marrow Transplant Program, Phoenix, Arizona
  - Myeloma Institute for Research and Therapy, University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope National Medical Center, Duarte, California
  - Cedars-Sinai, Los Angeles, California
  - University of California, Los Angeles, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana Blood and Marrow Transplantation Center, Beech Grove, Indiana
  - University of Iowa Hosptials and Clinics, Iowa City, Iowa
  - Fairview-University Medical Center, University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Kansas City Cancer Center, Kansas City, Missouri
  - Washington University School of Medicine, Division of Bone Marrow Transplantation and Leukemia, St Louis, Missouri
  - The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - St. Vincent's Comprehensive Cancer Center, New York, New York
  - New York Hospital, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - Utah Blood and Marrow Transplant Program, University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Vancouver General Hospital, Vancouver, British Columbia, Canada
- Universitätsklinikum Heidelberg,, Heidelberg, Germany

REFERENCES:
- [Result] DiPersio JF, Stadtmauer EA, Nademanee A, Micallef IN, Stiff PJ, Kaufman JL, Maziarz RT, Hosing C, Fruehauf S, Horwitz M, Cooper D, Bridger G, Calandra G; 3102 Investigators. Plerixafor and G-CSF versus placebo and G-CSF to mobilize hematopoietic stem cells for autologous stem cell transplantation in patients with multiple myeloma. Blood. 2009 Jun 4;113(23):5720-6. doi: 10.1182/blood-2008-08-174946. Epub 2009 Apr 10. PMID 19363221
- See also: Further information on multiple myeloma from the National Cancer Institute — http://www.nci.nih.gov/cancertopics/types/myeloma

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with multiple myeloma (MM) eligible for autologous hematopoietic stem cell transplant were recruited from 40 centers (38 in the U.S., 1 in Germany, 1 in Canada). The first participant was randomized on 04 February 2005 and the last participant's last study visit occurred on 22 January 2008. A total of 302 participants were randomized.
Groups:
- G-CSF Plus Plerixafor: Participants underwent mobilization with G-CSF for 4 days. On the evening of Day 4, participants received a dose of plerixafor. On each subsequent day, participants received a morning dose of G-CSF followed by apheresis and an evening dose of plerixafor for a maximum of 4 aphereses or until ≥ 6*10^6 CD34+ cells/kg were collected.
- G-CSF Plus Placebo: Participants underwent mobilization with G-CSF for 4 days. On the evening of Day 4, participants received a dose of placebo. On each subsequent day, participants received a morning dose of G-CSF followed by apheresis and an evening dose of placebo for a maximum of 4 aphereses or until ≥ 6*10^6 CD34+ cells/kg were collected.
Period: Overall Study
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Started | 148 | 154
Completed | 129 (1 participant was wrongly terminated due to 'other'; the participant stayed on study until death.) | 121 (1 participant was wrongly terminated due to 'other'; the participant stayed on study until death.)
Not Completed | 19 | 33
Not completed — Entered Rescue Procedure | 0 | 7
Not completed — Death | 7 | 7
Not completed — Elective Withdrawal | 5 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other | 6 | 9
Not completed — Failed mobilization | 0 | 4
Not completed — Intercurrent illness | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo | Total
Number analyzed (Participants) | 148 | 154 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (8.4) | 58.4 (8.6) | 58.3 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 47 | 95
  Male | 100 | 107 | 207
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 117 | 128 | 245
  African-American | 18 | 14 | 32
  Asian | 1 | 3 | 4
  Hispanic/Latino | 11 | 4 | 15
  Other | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Achieving a Target of ≥ 6*10^6 CD34+ Cells/kg in 2 or Fewer Days of Apheresis.
Description: Proportion of participants achieving a target of ≥ 6*10^6 CD34+ cells/kg in 2 or fewer days of apheresis. Central lab data were taken from Days 5 to 6 of the Treatment/Apheresis period. Each participant's value was calculated as the sum of all daily values collected over the 2 apheresis days.
Time Frame: up to Day 6
Population: Intent-to-Treat Population
Measure: Number; unit: proportion of participants
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Number analyzed (Participants) | 148 | 154
proportion of participants
  Proportion achieving target in ≤2 days | 0.716 | 0.344
  Proportion not achieving target in ≤2 days | 0.284 | 0.656

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with treatment emergent adverse events (AEs). The timeframe for treatment emergent AEs is defined as Day 1 (start of G-CSF Mobilization) to the day before starting chemotherapy (approximately 38 days later). AEs were reported regardless of relationship to study treatment. The investigator graded each AE using the World Health Organization (WHO) Adverse Event Grading Scale. AEs of Grade 3 were considered severe and Grade 4 were considered life-threatening.
Time Frame: up to Day 38
Population: Primary Safety population of all participants who received at least 1 mobilization dose of G-CSF or study treatment (plerixafor or placebo). Four participants did not receive G-CSF or any study treatment and were excluded from the safety analyses.
Measure: Number; unit: participants
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Number analyzed (Participants) | 147 | 151
participants
  Adverse Events (AEs) | 140 | 140
  Related AEs | 95 | 67
  AEs Leading to early treatment termination | 1 | 2
  AEs Leading to early termination | 3 | 0
  Grade 3 (severe) or 4 (life-threatening) AEs | 11 | 11
  Serious Adverse Events (SAEs) | 4 | 6

3. Secondary Outcome: Proportion of Participants Achieving a Target of ≥ 6*10^6 CD34+ Cells/kg in 4 or Fewer Days of Apheresis.
Description: Proportion of participants achieving a target of ≥ 6*10^6 CD34+ cells/kg in 4 or fewer days of apheresis. Central lab data were taken from Days 5 to 8 of the Treatment/Apheresis period. Each participant's value was calculated as the sum of all daily values collected over the 4 apheresis days.
Time Frame: up to Day 8
Population: Intent-to-Treat Population
Measure: Number; unit: proportion of participants
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Number analyzed (Participants) | 148 | 154
proportion of participants
  Proportion achieving target in ≤4 days | 0.757 | 0.513
  Proportion not achieving target in ≤4 days | 0.243 | 0.487

4. Secondary Outcome: Proportion of Participants Achieving a Target of ≥ 2*10^6 CD34+ Cells/kg in 4 or Fewer Days of Apheresis.
Description: Proportion of participants achieving a target of ≥ 2*10^6 CD34+ cells/kg in 4 or fewer days of apheresis. Central lab data were taken from Days 5 to 8 of the Treatment/Apheresis period. Each participant's value was calculated as the sum of all daily values collected over the 4 apheresis days.
Time Frame: up to Day 8
Population: Intent-to-Treat Population
Measure: Number; unit: proportion of participants
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Number analyzed (Participants) | 148 | 154
proportion of participants
  Proportion achieving target in ≤4 days | 0.953 | 0.883
  Proportion not achieving target in ≤4 days | 0.047 | 0.117

5. Secondary Outcome: Median Number of Days to ≥6*10^6 CD34+ Cells/kg
Description: The Kaplan Meier estimate of median number of days (number of days at which 50% of participants have experienced the event, accounting for censored values) in each treatment arm to collect an optimum number of cells (≥6*10^6 CD34+ cells/kg) for transplantation.
Time Frame: up to Day 8
Population: Intent-to-treat population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Number analyzed (Participants) | 144 | 150
Days | 1.0 [1.0 to 2.0] | 4.0 [2.0 to NA] — Not enough participants reached the threshold to support estimating the upper range.

6. Secondary Outcome: Median Number of Days to Polymorphonuclear (PMN) Cell Engraftment
Description: The Kaplan Meier estimate of median number of days to PMN engraftment (number of days at which 50% of participants have experienced the event, accounting for censored values) was a secondary efficacy endpoint. Engraftment was defined as PMN counts ≥ 0.5*10^9/L for 3 consecutive days or ≥ 1.0*10^9/L for 1 day. Time to engraftment corresponded to the first day that the criteria were met and was evaluated up to 12 months post transplant.
Time Frame: Up to Month 13
Population: Participants who received a stem cell transplant.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Number analyzed (Participants) | 142 | 136
Days | 11.0 [10.0 to 12.0] | 11.0 [11.0 to 12.0]

7. Secondary Outcome: Median Number of Days to Platelet (PLT) Engraftment
Description: The Kaplan Meier estimate of median number of days to PLT engraftment (number of days at which 50% of participants have experienced the event, accounting for censored values) was a secondary efficacy endpoint. Engraftment was defined as ≥ 20*10^9/L without transfusion for the preceding 7 days. Time to engraftment corresponded to the first day that the criteria were met and was evaluated up to 12 months post transplant.
Time Frame: Up to Month 13
Population: Participants who received a stem cell transplant
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Number analyzed (Participants) | 142 | 136
Days | 18.0 [16.0 to 22.0] | 18.0 [16.0 to 21.0]

8. Secondary Outcome: Graft Durability at 100 Days Post Transplantation
Description: The proportion of participants maintaining a durable graft at 100 days post-transplantation by at least 2 of the following criteria (without erythropoietin (EPO), G-CSF, or transfusions): (1) a platelet count >50000/µL without transfusion for at least 2 weeks, (2) hemoglobin >=10g/dL for at least 1 month, (3) and absolute neutrophil count >1000/µL for at least 1 week.
Time Frame: approximately Day 138
Population: Participants who received a stem cell transplant and were evaluable at 100 days post-transplant
Measure: Number; unit: proportion of participants
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Number analyzed (Participants) | 142 | 136
proportion of participants
  Proportion of participants with a durable graft | 0.986 | 0.978
  Proportion of participants without a durable graft | 0.014 | 0.022

9. Secondary Outcome: Graft Durability at 6 Months Post Transplantation
Description: The proportion of participants maintaining a durable graft at 6 months post-transplantation by at least 2 of the following criteria (without erythropoietin (EPO), G-CSF, or transfusions): (1) a platelet count >50000/µL without transfusion for at least 2 weeks, (2) hemoglobin >=10g/dL for at least 1 month, (3) and absolute neutrophil count >1000/µL for at least 1 week.
Time Frame: approximately Month 7
Population: Participants who received a stem cell transplant and were evaluable at 6 months post-transplant
Measure: Number; unit: proportion of participants
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Number analyzed (Participants) | 135 | 127
proportion of participants
  Proportion of participants with a durable graft | 0.985 | 0.984
  Proportion of participants without a durable graft | 0.015 | 0.016

10. Secondary Outcome: Graft Durability at 12 Months Post Transplantation
Description: The proportion of participants maintaining a durable graft at 12 months post-transplantation by at least 2 of the following criteria (without erythropoietin (EPO), G-CSF, or transfusions): (1) a platelet count >50000/µL without transfusion for at least 2 weeks, (2) hemoglobin >=10g/dL for at least 1 month, (3) and absolute neutrophil count >1000/µL for at least 1 week.
Time Frame: approximately Month 13
Population: Participants who received a stem cell transplant and were evaluable at 12 months post-transplant
Measure: Number; unit: proportion of participants
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Number analyzed (Participants) | 128 | 120
proportion of participants
  Proportion of participants with a durable graft | 0.992 | 0.992
  Proportion of participants without a durable graft | 0.008 | 0.008

ADVERSE EVENTS:
Time Frame: Day 1 (start of G-CSF Mobilization plus Treatment/Apheresis) to the day before starting chemotherapy. Chemotherapy typically started within 30 days of the last apheresis (which may have occurred on Day 5, 6, 7, or 8).
Description: Four participants did not receive any study treatment and were excluded from the safety analyses.
  In the event a participant experienced both a serious and a non-serious form of the same AE, they were included in the numerator of both AE tables. Each AE table includes all events, regardless of reported relationship to study treatment or grade.
Arm/Group | G-CSF Plus Plerixafor | G-CSF Plus Placebo
Serious Adverse Events (participants affected / at risk) | 4/147 | 6/151
Other Adverse Events (participants affected / at risk) | 140/147 | 140/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | G-CSF Plus Plerixafor (N=147) | G-CSF Plus Placebo (N=151)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Enterobacter bacteraemia (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Muscle spasticity (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | G-CSF Plus Plerixafor (N=147) | G-CSF Plus Placebo (N=151)
Anaemia (Blood and lymphatic system disorders) | 2 | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 4
Angina pectoris (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 2 | 4
Sinus tachycardia (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 4
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Eye irritation (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 5
Abdominal mass (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 4
Constipation (Gastrointestinal disorders) | 9 | 5
Dental discomfort (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 47 | 29
Dry mouth (Gastrointestinal disorders) | 6 | 6
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 1
Eructation (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 9 | 4
Frequent bowel movements (Gastrointestinal disorders) | 6 | 5
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 3 | 1
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 51 | 39
Oral soft tissue disorder (Gastrointestinal disorders) | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 11 | 13
Retching (Gastrointestinal disorders) | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 0
Tongue haematoma (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 17 | 9
Asthenia (General disorders) | 5 | 3
Catheter related complication (General disorders) | 1 | 5
Catheter site discharge (General disorders) | 1 | 1
Catheter site erythema (General disorders) | 1 | 4
Catheter site haematoma (General disorders) | 2 | 0
Catheter site haemorrhage (General disorders) | 6 | 6
Catheter site inflammation (General disorders) | 1 | 0
Catheter site oedema (General disorders) | 0 | 1
Catheter site pain (General disorders) | 14 | 19
Catheter site pruritus (General disorders) | 1 | 1
Catheter site related reaction (General disorders) | 7 | 4
Chest discomfort (General disorders) | 3 | 2
Chest pain (General disorders) | 2 | 2
Chills (General disorders) | 4 | 4
Discomfort (General disorders) | 0 | 1
Fatigue (General disorders) | 40 | 41
Feeling abnormal (General disorders) | 0 | 1
Feeling cold (General disorders) | 2 | 2
Feeling hot (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Influenza like illness (General disorders) | 3 | 1
Infusion site mass (General disorders) | 1 | 0
Infusion site thrombosis (General disorders) | 0 | 1
Injection site bruising (General disorders) | 3 | 2
Injection site discharge (General disorders) | 1 | 0
Injection site erythema (General disorders) | 32 | 5
Injection site haemorrhage (General disorders) | 4 | 1
Injection site induration (General disorders) | 1 | 0
Injection site irritation (General disorders) | 3 | 3
Injection site pain (General disorders) | 3 | 1
Injection site paraesthesia (General disorders) | 1 | 0
Injection site pruritus (General disorders) | 5 | 1
Injection site rash (General disorders) | 2 | 0
Injection site reaction (General disorders) | 1 | 0
Injection site swelling (General disorders) | 1 | 1
Irritability (General disorders) | 1 | 0
Malaise (General disorders) | 5 | 1
Mucosal inflammation (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 12 | 10
Pain (General disorders) | 11 | 11
Peripheral coldness (General disorders) | 0 | 1
Pitting oedema (General disorders) | 0 | 1
Pyrexia (General disorders) | 8 | 11
Sensation of pressure (General disorders) | 0 | 1
Vessel puncture site haematoma (General disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Tinea manuum (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 4
Urinary tract infection (Infections and infestations) | 0 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Citrate toxicity (Injury, poisoning and procedural complications) | 6 | 4
Contusion (Injury, poisoning and procedural complications) | 4 | 5
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypertension (Injury, poisoning and procedural complications) | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Tooth injury (Injury, poisoning and procedural complications) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 3
Blood calcium decreased (Investigations) | 0 | 1
Blood glucose decreased (Investigations) | 0 | 1
Blood magnesium decreased (Investigations) | 1 | 1
Blood potassium decreased (Investigations) | 2 | 1
Blood pressure increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 6 | 6
Body temperature increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Cardiac murmur (Investigations) | 1 | 0
Culture positive (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 0 | 1
Heart rate irregular (Investigations) | 1 | 4
Lymph node palpable (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 6 | 6
Decreased appetite (Metabolism and nutrition disorders) | 6 | 5
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 19 | 29
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 | 16
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Tetany (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 34
Bone pain (Musculoskeletal and connective tissue disorders) | 53 | 64
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Jaw disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 8
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 | 5
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 5
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 11
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lentigo (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 1
Burning sensation (Nervous system disorders) | 1 | 0
Coordination abnormal (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 17 | 10
Dysgeusia (Nervous system disorders) | 7 | 2
Dyskinesia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 30 | 35
Hypoaesthesia (Nervous system disorders) | 8 | 7
Lethargy (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 33 | 34
Parosmia (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 2 | 2
Sensory disturbance (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 3 | 3
Abnormal dreams (Psychiatric disorders) | 0 | 1
Anticipatory anxiety (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 9 | 6
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Emotional distress (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 10 | 11
Restlessness (Psychiatric disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 2
Nocturia (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Vaginal pain (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Ephelides (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 5
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 5 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 4 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Scar (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 4 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 2 | 1
Hot flush (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 2 | 5
Hypotension (Vascular disorders) | 2 | 5
Orthostatic hypotension (Vascular disorders) | 1 | 0
Pallor (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.